CLINICAL TRIAL: NCT02124408
Title: Mobile Phone Personalized Intervention for Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ningbo Beilun District Traditional Chinese Medicine Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: H20132175
Record Dates: First submitted 2014-04-19; First posted 2014-04-28 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Intervention group (Experimental): Personalized Behavioral Intervention
  Interventions: Behavioral: Personalized Behavioral Intervention
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Personalized Behavioral Intervention
  Arms: Intervention group

SUMMARY:
With the development of economy and change of lifestyles, it is characterized that there is a dramatic increase of diabetes in China. Changes in lifestyle/self-care behaviors by diabetes patients are required to improve blood glucose and subsequent outcomes. Mobile phone intervention was a kind of high cost efficiency and high quality health care. Our study evaluated a diabetes coaching system, using mobile phones and patient/provider portals for patient-specific treatment and communication.

ELIGIBILITY:
Inclusion Criteria:

1. Physician diagnosis of type 2 diabetes
2. Age 20 years and more
3. The local resident

Exclusion Criteria:

1. Not currently managed by study physicians
2. Pregnant
3. Active substance, alcohol, or drug abuser
4. Psychotic or schizophrenic under activecare
5. Severe hearing or visual impairment
6. No telephone or mobile phone

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
change in glycated hemoglobin levels | baseline and 6 months
  Blood sample would be collected and HbA1C level would be assessed in baseline and 6 months later.Change in glycated hemoglobin levels will be compared between the two group.

SECONDARY OUTCOMES:
changes in patient-reported diabetes symptoms | baseline and 6 months
  Diabetes symptoms such as polydipsia, polyuria and polyphagia of all participants would be obtained by questionnaire in baseline and 6 months and compared between the two groups.
control of diabetic complications | baseline and 6 months
  Blood pressure, blood lipid, weight and sleep quality etc.would be obtained by physical or lab examination or questionnaire in baseline and 6 months. The percentage of patients with well-control of blood pressure (BP≤130/80mmHg),weight (BMI≤24kg/m2) and sleep quality(PSQI score≤5) etc.will be compared between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo Beilun District Traditional Chinese Medicine Hospital, Ningbo, Zhejiang, China